CLINICAL TRIAL: NCT05090254
Title: The Effect of Perioperative Cardiac Output-guided Goal-directed Hemodynamic Therapy (GDT) on Perioperative Oxygen Delivery, Consumption, and Microcirculatory Perfusion in Comparison to Routine Hemodynamic Management
Brief Title: The Effect of Perioperative Cardiac Output-guided GDT on Oxygen Delivery, Consumption, and Microcirculatory Perfusion
Acronym: CUSTOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-10141-BO-ff
Record Dates: First submitted 2021-08-29; First posted 2021-10-22 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Caridac Output-guided Goal-directed Hemodynamic Therapy; Oxygen Delivery; Oxygen Consumption; Microcirculatory Perfusion; Major Non-cardiac Surgery; Postoperative Acute Kidney Injury; Postoperative Acute Myocardial Injury
Keywords: non-cardiac surgery; oxygen consumption; oxygen delivery; microcirculatory perfusion; goal-directed hemodynamic therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cardiac output maximization group (Active Comparator): Patients will be treated according to a goal-directed therapy protocol aiming at a cardiac output maximization.
  Detailed protocol adapted from Edwards, M.R., et al., Optimisation of Perioperative Cardiovascular Management to Improve Surgical Outcome II (OPTIMISE II) trial: study protocol for a multicentre international trial of cardiac output-guided fluid therapy with low-dose inotrope infusion compared with usual care in patients undergoing major elective gastrointestinal surgery. BMJ Open, 2019. 9(1): p. e023455.
  Interventions: Other: Treatment algorithms targeting cardiac output
- Cardiac output personalization group (Active Comparator): Patients will be treated according to a goal-directed therapy protocol aiming at a personalized cardiac output goal determined with preoperative cardiac output assessment.
  Detailed protocol adapted from Nicklas, J.Y., et al., Personalised haemodynamic management targeting baseline cardiac index in high-risk patients undergoing major abdominal surgery: a randomised single-centre clinical trial. Br J Anaesth, 2020. 125(2): p. 122-132.
  Interventions: Other: Treatment algorithms targeting cardiac output
- Routine management group (No Intervention): Patients will be treated according to routine hemodynamic management.

INTERVENTIONS:
Other: Treatment algorithms targeting cardiac output — Treatment algorithms targeting maximization or personalization of cardiac output
  Arms: Cardiac output maximization group; Cardiac output personalization group

SUMMARY:
Perioperative cardiac output-guided goal-directed therapy (GDT) triggers fluid, vasopressor, and inotrope administration assuming that optimizing cardiac output (i.e., global blood flow) ensures adequate oxygen delivery and microcirculatory perfusion - that are usually not directly monitored during goal-directed therapy. There is increasing evidence that perioperative cardiac output-guided goal-directed therapy may reduce postoperative complications compared to routine hemodynamic management in high-risk patients having major surgery. The effect of cardiac output-guided goal-directed therapy algorithms on perioperative oxygen delivery and consumption as well as microcirculatory perfusion, however, is unknown.

The investigators aim to investigate the effect of using different cardiac output-guided goal-directed therapy algorithms on perioperative oxygen delivery and consumption as well as sublingual microcirculatory perfusion compared to routine perioperative hemodynamic management in patients having major abdominal surgery with general anesthesia.

DETAILED DESCRIPTION:
Perioperative cardiac output-guided goal-directed therapy (GDT) triggers fluid, vasopressor, and inotrope administration assuming that optimizing cardiac output (i.e., global blood flow) ensures adequate oxygen delivery and microcirculatory perfusion - that are usually not directly monitored during goal-directed therapy. There is increasing evidence that perioperative cardiac output-guided goal-directed therapy may reduce postoperative complications compared to routine hemodynamic management in high-risk patients having major surgery. The effect of cardiac output-guided goal-directed therapy algorithms on perioperative oxygen delivery and consumption as well as microcirculatory perfusion, however, is unknown.

With technological advancements a distinct monitoring of oxygen delivery and consumption as well as microcirculatory perfusion in the perioperative period has become possible. Using new technologies, a detailed understanding of the effect of cardiac output-guided goal-directed therapy on perioperative oxygen delivery and consumption as well as microcirculatory perfusion is of vital importance to further develop and improve perioperative hemodynamic treatment strategies.

In this pilot randomized-controlled trial, the investigators therefore aim to investigate the effect of using different cardiac output-guided goal-directed therapy algorithms on perioperative oxygen delivery and consumption as well as sublingual microcirculatory perfusion compared to routine perioperative hemodynamic management in patients having major abdominal surgery with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) having elective major abdominal surgery with general anesthesia
* Expected duration of surgery at least 120 minutes
* Planned postoperative monitoring in intensive care unit

Exclusion Criteria:

* Emergency surgery
* Age <18 years
* Body weight <50 kg
* Pregnancy
* Atrial fibrillation
* Planned patient positioning in other position than supine position
* Surgery within the last 30 days
* Inaccessibility of the head during surgery
* Peripheral artery disease stage ≥IIb
* Chronic vasculitis
* Supraglottic airway management
* Enterostomy repair surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Perioperative changes in oxygen delivery | after induction of general anesthesia, during the last 30 minutes of surgery, within 6 hours after surgery, day 1, 2, 3 after surgery
  assessed via blood gas analysis
Perioperative changes in oxygen consumption | baseline awake, after induction of general anesthesia, during the last 30 minutes of surgery, within 6 hours after surgery, day 1, 2, 3 after surgery
  assessed via indirect calorimetry

SECONDARY OUTCOMES:
Perioperative changes of microcirculation | baseline awake, after induction of general anesthesia, during the last 30 minutes of surgery, within 6 hours after surgery, day 1, 2, 3 after surgery
  assessed via Incident Darkfield technology
Perioperative changes in cardiac output | baseline awake, after induction of general anesthesia, during the last 30 minutes of surgery, within 6 hours after surgery, day 1, 2, 3 after surgery
  assessed via pulse wave analysis

OTHER OUTCOMES:
Incidence of postoperative myocardial injury | baseline awake, within 6 hours after surgery, and on day 1, 2, and 3 after surgery
  assessed via blood samples
Incidence of acute kidney injury | baseline awake, within 6 hours after surgery, and on day 1, 2, and 3 after surgery
  assessed via blood samples
Perioperative changes in urethral perfusion index | after induction of general anesthesia, during the last 30 minutes of surgery, within 6 hours after surgery, day 1, 2, 3 after surgery
  assessed via urethral photoplethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Saugel, Prof., MD, Principal Investigator — The University Medical Center Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany